CLINICAL TRIAL: NCT03145337
Title: A Prospective, Randomized, Multi-Center Clinical Study Comparing Outcomes in Patients Undergoing Prosthetic, Acellular Dermal Matrix (ADM) Assisted, Immediate Post-Mastectomy Breast Reconstruction
Brief Title: Reconstruction Outcomes in Immediate Post-mastectomy Breast Reconstruction With ADM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Musculoskeletal Transplant Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MTF 16-04-01
Record Dates: First submitted 2017-05-03; First posted 2017-05-09 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-05

CONDITIONS: Breast Reconstruction

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled
Who Masked: Outcomes Assessor
Masking Description: 3-4 independent breast surgeons using predefined criteria will assess the aesthetic outcomes of each subject using photographs of their pre-mastectomy and 12 month post-reconstructions. The surgeons will not be apprised of the ADM type or post-mastectomy site/surgeon
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Active Comparator): FlexHD ADM
  Interventions: Biological: FlexHD ADM (Cohort A)
- Cohort B (Active Comparator): AlloDerm RTU ADM
  Interventions: Biological: AlloDerm RTU ADM (Cohort B)

INTERVENTIONS:
Biological: FlexHD ADM (Cohort A) — Tissue assisted breast reconstruction with FlexHD pliable perforated ADM
  Other Names: FlexHD ADM
  Arms: Cohort A
Biological: AlloDerm RTU ADM (Cohort B) — Tissue assisted breast reconstruction with AlloDerm RTU perforated ADM
  Other Names: AlloDerm RTU ADM
  Arms: Cohort B

SUMMARY:
Evaluation and comparison of clinical and aesthetic outcomes associated with the use of two allograft dermal matrices (ADMs) currently in use for tissue assisted immediate post-mastectomy breast reconstruction.

DETAILED DESCRIPTION:
This is a level one, prospective, randomized, controlled multi-center clinical study comparing two types of acellular dermal matrices (ADMs) currently used in immediate post-mastectomy prosthetic breast reconstruction. Comparison of these two ADMs will be made in the areas of reconstructive clinical outcomes and aesthetic outcomes. Patients will be randomized into one of two ADM groups as part of their immediate post-mastectomy breast reconstruction. Patients in both groups will be followed for twelve months after their reconstructive surgery. Clinical outcomes will be documented at 1 month, 3 months, 6 months and 12 months following breast reconstructive surgery. For one-stage breast reconstruction, aesthetic outcomes will be assessed and documented at 6 and 12 months following implant placement. For two-stage reconstruction, patients will be evaluated for aesthetic outcomes at a time point 6-12 months following expander-to-implant exchange if it does not coincide with the 12 month post-mastectomy visit.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled to undergo immediate, post-mastectomy, tissue assisted breast reconstruction, Reconstruction shall be either one-stage (direct-to-implant) or two-stage, unilateral or bilateral, prophylactic or therapeutic
2. Females at least 18 years of age
3. Non-smokers, former smokers and/or smokers who have not smoked within 1 month before surgery, and who agree to not smoke or utilize e-cigarettes during the post-operative period
4. Have signed a written informed consent
5. Have the ability to understand and comply with the requirements and follow-up time points of the study

Exclusion Criteria:

1. Previous breast surgery with the exception of biopsy
2. Previous radiation treatment in either breast at any time
3. Undergoing autologous breast reconstruction
4. Pre-pectoral implant placement
5. Undergoing delayed reconstruction
6. Requiring Wise pattern reduction of mastectomy skin flap
7. History of chronic steroid use within the past 6 months
8. History of HIV positive
9. Previous organ transplant
10. Pregnant or lactating females
11. Clinically significant systemic disease, as determined by the investigator, which could affect study participation or study results

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Post Reconstruction Complication Rates | 12 months
  To compare the overall complication rate between the cohorts defined as either 1) post-operative infection specific to the reconstructed breast(s) requiring either intravenous antibiotic treatment or operative intervention, 2) seroma, and/or 3) reconstructive failure

SECONDARY OUTCOMES:
Comparison of Each Complication Rate | 12 months
  To compare each complication rate between the cohorts defined as 1) post-operative infection specific to the reconstructed breast(s) requiring either intravenous antibiotic treatment or operative intervention 20 seroma 3) reconstructive failure and 4) reoperation for reasons other than infection
Comparison of Aesthetic Outcomes (Photographs) | 12 months
  A blinded comparison of aesthetic outcomes (photographs) using pre-defined criteria

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Northwestern University Medical Center, Chicago, Illinois
  - NorthShore Health Systems, Evanston, Illinois
  - Louisiana State Health Science Center, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Faulkner Brigham & Women's Hospital, Jamaica Plain, Massachusetts
  - New York University Langone Medical Center, New York, New York
  - Harris Methodist Southlake Hospital, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: No